CLINICAL TRIAL: NCT03931954
Title: PREPARE STUDY: PRevalence of the Eosinophilic Phenotype Among SeveRE Asthma Patients in AstraZeneca International Region. A Multinational, Cross-Sectional, Multicenter Study
Brief Title: Prevalence of the Eosinophilic Phenotype Among Severe Asthma Patients
Acronym: PREPARE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D2287R00140
Record Dates: First submitted 2019-04-10; First posted 2019-04-30 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Severe Asthma
Keywords: eosinophilic asthma; severe asthma; prevalence; phenotype; atopic phenotype; eosinophilic phenotype
MeSH Terms: conditions — Asthma; Pulmonary Eosinophilia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study population: Patients completing the inclusión criteria

SUMMARY:
The purpose of this cross-sectional, multicenter study is to determine the prevalence of an eosinophilic phenotype of blood eosinophil count ≥ 300 cells/mm3 among severe asthma patients who attend to sites specialized in the management of severe asthma in several countries in the AstraZeneca International Region. The prevalence of an atopic phenotype and asthma control, will also be studied.

DETAILED DESCRIPTION:
To determine the prevalence of an eosinophilic phenotype of blood eosinophil count ≥ 300 cells/mm3 among severe asthma patients attending their routine clinical visit at sites specialized in the management of severe asthma in several countries in the AstraZeneca International Region. The prevalence of an atopic phenotype and the status of asthma control, will also be studied. It is expected that this study will contribute to the understanding of severe asthma, ultimately helping to inform therapeutic decisions and addressing patients' needs.

ELIGIBILITY:
Inclusion Criteria

Patients must fulfil all of the following inclusion criteria to be included in the study:

* Male or female patient, aged 12 years or older by the time of study entry
* Patient visiting a participating center for a routine clinical appointment
* Patient is willing and able to provide a blood sample for IgE and eosinophil levels determination as part of their routine clinical visit
* Diagnosis of severe asthma for at least one year as defined by:
* Treatment with guidelines-suggested medications for Global Initiative for Asthma (3) steps 4-5 asthma
* Patients or their legal guardian, who voluntarily sign and date the informed consent form prior to study entry.

Exclusion Criteria

* Patients with a diagnosis of chronic obstructive pulmonary disease or other chronic respiratory condition beyond severe asthma
* An acute or chronic condition that, in the investigator's opinion, would limit the patient's ability to participate in this study Patients who are currently under a biologic therapy to treat their severe asthma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include patients from 12 years and older with severe asthma, as per the definition of the GINA 2018 Guidelines (GINA, 2018). Patients will be identified and invited to participate in the study consecutively, as they attend their routine clinical visit at the research centers.
  To be included in the study, each patient should meet all the inclusion criteria and none of the exclusion criteria described in the sections below. Patients should provide written, informed consent prior to any study-specific procedures.
  The enrolment period will be approximately 8 months or until the required number of patients has been included, whichever occurs first
Sampling Method: Non-Probability Sample
Enrollment: 794 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-11-26 (Actual); Study Completion 2020-11-26 (Actual)

PRIMARY OUTCOMES:
Blood Eosinophil count | There is only one study visit. During that study visit the sample will be collected
  The level of eosinophils in the blood will be assessed from this blood sample and reported
Total serum IgE | There is only one study visit. during that visit the sample will be collected
  Total serum IgE will be assessed from this blood sample and reported

CONTACTS AND LOCATIONS:
Overall Officials: Maarten beekman, MD, Study Chair — medical lead respiratory International; Monica Olmos, MD, Study Chair — Study delivery lead
Locations (17):
- Argentina (2):
  - Research Site, Buenos Aires
  - Research Site, Rosario
- Chile (2):
  - Research Site, Curicó
  - Research Site, Santiago
- Colombia (4):
  - Research Site, Barranquilla
  - Research Site, Bogotá
  - Research Site, Bucaramanga
  - Research Site, Pereira
- Research Site, San José, Costa Rica
- Mexico (5):
  - Research Site, Guadalajara
  - Research Site, Mérida
  - Research Site, Puebla City
  - Research Site, San Juan del Río
  - Research Site, Villahermosa
- Saudi Arabia (3):
  - Research Site, Dammam
  - Research Site, Jeddah
  - Research Site, Riyadh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Al-Jahdali H, Wali S, Albanna AS, Allehebi R, Al-Matar H, Fattouh M, Beekman M. Prevalence of eosinophilic, atopic, and overlap phenotypes among patients with severe asthma in Saudi Arabia: a cross-sectional study. BMC Pulm Med. 2022 Feb 17;22(1):67. doi: 10.1186/s12890-022-01856-9. PMID 35177038
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D2287R00140&attachmentIdentifier=706cb728-2854-4287-a5b9-0d84bcd0a71c&fileName=CSR_PREPARE_V_0.5_CTT_with_Milestones_Combined.pdf&versionIdentifier=